CLINICAL TRIAL: NCT06709417
Title: A Phase II Clinical Study of Sintilimab Combined with Chemotherapy Followed by Concurrent Chemoradiotherapy for Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma (ESCC) (NICE-CS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jun Liu, associate professor, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICE-CS
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab; Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): Eligible participants will first receive two cycles of sintilimab in combination with liposomal paclitaxel and cisplatin. After two cycles, an evaluation will be conducted. Patients deemed eligible for surgery will undergo surgical resection, followed by up to one year of adjuvant sintilimab. The necessity of postoperative adjuvant radiotherapy will be determined by the investigator.
  For patients deemed ineligible for surgery, concurrent chemoradiotherapy will be administered. Four weeks after the completion of concurrent chemoradiotherapy, a second surgical evaluation will be performed. Patients eligible for surgery at this stage will undergo surgical resection followed by adjuvant sintilimab treatment. Those who remain ineligible for surgery will continue sintilimab treatment after concurrent chemoradiotherapy.
  Interventions: Drug: Sintilimab; Drug: Chemotherapy; Radiation: radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg iv Q3W
Drug: Chemotherapy — Liposomal paclitaxel: 150mg/m2, Q3W + cisplatin: 75mg/m2, Q3W (combined with PD-1 therapy) Liposomal paclitaxel: 50mg/m2, Q3W + cisplatin: 20mg/m2, Q3W (combined with radiotherapy )
Radiation: radiotherapy — The total dose is 5040cCy in 28 fractions (5 days per week, 1.8 Gy/day).

SUMMARY:
This is a prospective, single-arm, phase II clinical study designed to evaluate the efficacy and safety of sintilimab combined with chemotherapy, followed by sequential concurrent chemoradiotherapy as conversion therapy, in treatment-naïve esophageal squamous cell carcinoma (ESCC) patients with cT4bN-/+M0 and/or cTanyN+M0 staging (including those with extracapsular invasion of mediastinal lymph nodes).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to the initiation of any study-related procedures.
2. Age: ≥20 years and ≤75 years, no gender restrictions.
3. Diagnosed with esophageal squamous cell carcinoma (ESCC) based on histopathology and imaging, with clinical staging of cT4bN-/+M0 and/or cTanyN+M0 (extracapsular invasion of mediastinal lymph nodes).
4. Thoracic segment esophageal squamous cell carcinoma.
5. Primary lesion is inoperable or inoperable due to extracapsular invasion of mediastinal lymph nodes.
6. ECOG performance status (PS) of 0-1.
7. Estimated survival time ≥6 months.
8. No prior antitumor therapy for esophageal cancer, including but not limited to chemotherapy, radiotherapy, targeted therapy, or immunotherapy.
9. At least one measurable lesion as per RECIST 1.1 criteria.
10. No surgical contraindications based on preoperative evaluation of organ function.
11. Adequate organ function
12. Female participants of childbearing potential must have a negative urine or serum pregnancy test within three days prior to receiving the first dose of study medication (Cycle 1, Day 1). If the urine pregnancy test result is inconclusive, a serum pregnancy test is required. Non-childbearing potential is defined as postmenopausal for at least one year, surgical sterilization, or hysterectomy.

Participants of childbearing potential (male or female) must use highly effective contraception methods (with an annual failure rate <1%) throughout the study and for 120 days after the last dose of the investigational drug or 180 days after the last dose of chemotherapy, whichever is longer.

Exclusion Criteria:

1. Diagnosis of malignancies other than esophageal cancer within 5 years prior to the first dose of the investigational drug (excluding radically treated basal cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the lung, or T1a non-invasive adenocarcinoma).
2. Patients with existing or high-risk tracheoesophageal or aortoesophageal fistulas.
3. Presence of distant metastases.
4. Current participation in an interventional clinical study or receipt of other investigational drugs or devices within 4 weeks prior to the first dose.
5. Prior treatment with anti-PD-1, anti-PD-L1, or any other agents targeting stimulatory or co-inhibitory T-cell receptors (e.g., CTLA-4, OX-40, CD137).
6. Receipt of systemic antitumor traditional Chinese medicine or immunomodulatory drugs (including thymosin, interferon, or interleukin) within 2 weeks prior to the first dose, except for local use to control pleural effusion.
7. Active autoimmune disease requiring systemic therapy (e.g., disease-modifying agents, corticosteroids, or immunosuppressive drugs) within 2 years prior to the first dose, excluding replacement therapy (e.g., thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency).
8. Use of systemic corticosteroids (excluding nasal, inhaled, or other locally administered corticosteroids) or other immunosuppressive drugs within 7 days prior to the first dose, except for physiological doses of corticosteroids (≤10 mg/day prednisone or equivalent).
9. History of allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
10. Known hypersensitivity to active ingredients or excipients in the investigational product.
11. Failure to recover adequately (≤Grade 1 or baseline) from prior therapy-induced toxicities and/or complications prior to initiating treatment (excluding fatigue or alopecia).
12. Known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive).
13. Untreated active hepatitis B, defined as HBsAg positivity with HBV DNA levels exceeding the upper limit of normal (ULN) at the study center. Subjects meeting the following criteria are eligible: HBV DNA <1000 copies/mL (200 IU/mL) prior to the first dose and on antiviral therapy during chemotherapy to prevent reactivation. Subjects with anti-HBc(+), HBsAg(-), anti-HBs(-), and negative HBV DNA do not require prophylactic antiviral therapy but need close monitoring for reactivation.
14. Active hepatitis C infection, defined as HCV antibody positivity and HCV RNA levels above the lower limit of detection.
15. Receipt of live vaccines within 30 days prior to the first dose (Cycle 1, Day 1), except for injectable inactivated influenza vaccines administered within 30 days prior to the first dose. Intranasal attenuated live influenza vaccines are not allowed.
16. Pregnant or breastfeeding women.
17. History of gastrointestinal bleeding within 6 months prior to treatment or concurrent coagulation disorders, or patients on thrombolytic or anticoagulant therapy with a high risk of bleeding.
18. Any severe or uncontrolled systemic disease, including but not limited to:

    1. Major, symptomatic, and poorly controlled abnormalities in cardiac rhythm, conduction, or morphology on resting ECG, such as complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmias, or atrial fibrillation.
    2. Unstable angina or congestive heart failure classified as NYHA grade ≥2.
    3. Arterial thrombosis, embolism, or ischemia within 6 months prior to enrollment, including myocardial infarction, unstable angina, cerebrovascular accidents, or transient ischemic attacks.
    4. Poorly controlled blood pressure (systolic BP >140 mmHg, diastolic BP >90 mmHg).
    5. History of non-infectious pneumonitis requiring corticosteroid therapy within 1 year prior to the first dose or current clinically active interstitial lung disease.
    6. Active pulmonary tuberculosis.
    7. Active or uncontrolled infections requiring systemic therapy.
    8. Clinically active diverticulitis, intra-abdominal abscess, or gastrointestinal obstruction.
    9. Liver diseases, such as cirrhosis, decompensated liver disease, or acute/chronic active hepatitis.
    10. Poorly controlled diabetes mellitus (fasting blood glucose >10 mmol/L).
    11. Proteinuria ≥++ on urinalysis, confirmed by 24-hour urinary protein quantification >1.0 g.
    12. Psychiatric disorders that interfere with compliance or treatment.
19. Any history, evidence of disease, abnormal treatment, or laboratory findings that could interfere with study outcomes, impede full participation, or, in the investigator's opinion, render the subject unsuitable for the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-yr OS rate | 24 months
  The percentage of people in the study who are alive two years after the start of treatment.

SECONDARY OUTCOMES:
R0 resection rate | 24 months
  The proportion of R0 resections achieved during surgery.
pCR rate | 24 months
  pathological complete response (pCR) is defined as no viable residual tumor.
MPR rate | 24 months
  The proportion of patients achieved MPR. The major pathologic response (MPR) is defined as residual viable tumor of less than or equal to 10%.
EFS | 24 months
  Refers to the time from the start of treatment to the first occurrence of any of the following events: disease progression that is inoperable, local or distant recurrence, death due to any cause, etc.
OS | 24 months
  The time from the start of treatment to the death of the subject due to various causes.
surgical conversion rate | 24 months
  The proportion of participants assessed as eligible for surgical resection after treatment among the total number of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No